CLINICAL TRIAL: NCT06731816
Title: The Comparison of the Effects of Neck Exercises With or Without the Stabilization Exercises on Pain, Posture, and Sleep Quality in Office Workers With Neck Pain
Brief Title: The Effect of Stabilization Exercises on Pain, Posture, and Sleep in Office Workers With Neck Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Seda BAKTIR, Assist. Prof, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LHU-FTR-ZSBD-02
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain; Neck Pain Treatment
Keywords: Sleep Quality; Posture; Pain; Neckache; Neck Pains; Exercise; Neck Exercises; Stabilization Exercises
MeSH Terms: conditions — Neck Pain; Sleep Initiation and Maintenance Disorders; Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel group comparison
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neck and stabilization exercise group (Active Comparator): In addition to neck stretching, range of motion, and isometric exercises, spinal stabilization exercises will be applied.
  Interventions: Other: Neck and stabilization exercise group
- Neck exercise group (Active Comparator): Neck stretching, range of motion, and isometric exercises will be applied.
  Interventions: Other: Neck exercise group

INTERVENTIONS:
Other: Neck and stabilization exercise group — Participants in this group will attend 2 sessions per week for 8 weeks, for a total of 16 sessions. In addition to neck stretching, range of motion, and isometric exercises applied in the neck exercise group, they will also apply spinal and cervical region stabilization exercises.
  Arms: Neck and stabilization exercise group
Other: Neck exercise group — Participants in this group will attend 2 sessions per week for 8 weeks, for a total of 16 sessions. They will perform neck stretching, range of motion and isometric exercises.
  Arms: Neck exercise group

SUMMARY:
With this study that will be examined the effects of stabilization exercises applied in addition to neck exercises on neck pain, posture and sleep quality in office workers with neck pain.

DETAILED DESCRIPTION:
Today, technological devices play a significant role in both professional and personal aspects of our lives. While computer use in office workers increases work productivity, it also brings about certain health risks by affecting posture and the musculoskeletal system. During screen use, the repetitive and prolonged forward movement of the head and arms results in a kyphotic posture and an increased neck flexion angle, which causes pain in the cervical region. When the head is in a neutral position, the amount of load carried by the cervical region is estimated to be around 4.5-5.5 kg, whereas with a 15° neck flexion, this load increases to 12.25 kg, and with a 30° flexion angle, it reaches approximately 13.61 kg. Increased flexion angles in the cervical region lead to an increase in mechanical stress on ligaments, tendons, muscles, and bones, and this stress poses a potential risk for the development of arthritis, disc degeneration, and headaches.

Musculoskeletal disorders caused by these symptoms are believed to reduce work productivity and lead to employees taking breaks from their tasks. Prolonged use of smartphones or computers is associated with increased anxiety and stress levels, as well as sleep problems. Pilates has become an increasingly popular form of exercise in the rehabilitation field in recent years. Joseph Pilates referred to the core region as the "powerhouse" and considered core control to be a fundamental component of body movement. According to Pilates, learning to properly engage the core muscles improves movement quality, enhances posture, and provides better stabilization. Exercises targeting the deep stabilizing muscles strengthen the torso, correct posture, and improve balance.

Pilates training plays a role in increasing strength and endurance, restoring normal proprioceptive mechanisms, and maintaining flexibility. For this reason, it is recommended in both preventive and therapeutic exercise programs. The aim of this study is to create two different exercise programs for office workers with neck pain and to investigate the effects of stabilization exercises, applied in addition to neck exercises, on neck pain, posture, and sleep quality.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria for the Study:

* Volunteering to participate in the study and approving the informed consent form,
* Using a computer, tablet and/or phone for more than 3 hours per day for the last 6 months,
* Having recurrent or persistent pain in the neck region for at least 3 months,
* Having a Neck Disability Scale score of 15 points or higher,
* Having a VAS Pain score of 5 or higher.

Exclusion Criteria:

* Having a neurological diagnosis,
* Having a radiologically confirmed orthopedic diagnosis from the neck region (neck hernia, fracture, dislocation, spondylolisthesis),
* Having a systemic and chronic disease diagnosis that can affect the neck region and joints,
* Having a history of surgical intervention or trauma from the neck region,
* Having cognitive impairment that makes communication and evaluation difficult.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 8 weeks
  This scale consists of a horizontal line 10 cm (100mm) in length, where the starting point marked as 0 represents "no pain," and the point marked as 10 represents "the most intense pain." Participants are asked to mark the point on this line that corresponds to their current level of pain.
Neck Disability Index (NDI) | 8 weeks
  Neck Disability Index is a commonly used self-reported questionnaire designed to assess the level of disability caused by neck pain. It evaluates how neck pain affects a person's daily activities, including their ability to work, engage in physical activities, and manage personal care. The NDI consists of 10 sections, each with a set of questions that cover different aspects of daily life, such as pain intensity, personal care, lifting, reading, headaches, concentration, sleeping, driving, and working. Each section is scored from 0 to 5, with higher scores indicating greater disability. A total score between 15 and 24 indicates moderate disability, a score between 25 and 34 indicates severe disability, and a score of 35 or above indicates complete disability.
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  Pittsburgh Sleep Quality Index is a widely used tool for assessing sleep quality and disturbances. It is a self-reported questionnaire that evaluates various aspects of sleep over a one-month period. The PSQI consists of 19 items grouped into seven components, each assessing a different aspect of sleep. Each component is scored from 0 to 3, with higher scores indicating worse sleep quality or greater disturbances. The total score is calculated by adding the component scores, with a maximum possible score of 21. A total score above 5 is typically considered indicative of poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Z.Seda Baktir Dogan Assist Profesor, Doctorate, Principal Investigator — Lokman Hekim University
Locations (1):
- Lokman Hekim University Health Sciences Institute, Ankara, Çankaya/Sögütözü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the beginning of the study, it is more suitable to share. Yet, it is early to estimate the progression of study.